CLINICAL TRIAL: NCT05896111
Title: Effect of Whole Body Vibration on Upper Limb Range of Motion and Strength in Children With Hemiparetic Cerebral Palsy
Brief Title: Whole Body Vibration for Hemiparetic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Haytham Ibrahim Morsi, Senior., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.1993
Record Dates: First submitted 2023-05-27; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Physical Therapy
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: pilot testing to get sample.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- designed physiotherapy program (Experimental): These exercises included:
  Passive stretching exercises for elbow and wrist flexors. Weight-bearing exercises for the upper limbs. Stimulation of the protective reactions of the upper limbs in all directions. Strengthening exercises for antagonists of the spastic muscles, including elbow and wrist extensors, using different toys and motivation to encourage the children to perform the desired exercises (El-shamy, 2018).
  The treatment session for 1hour 5 days / week for 4 weeks.
  Interventions: Procedure: Physical therapy exercises.
- Whole body vibration. (Experimental): Each child will be seated on an armless chair in front of the platform and instructed to flex both shoulders at 90°, slightly bend both elbows, and then bend the trunk forward to allow both hands to be placed on the platform. Each subject will be allowed to hold the palms slightly off the platform to minimize discomfort and prevent strong stimulation of the organs, eyes, and head.
  Interventions: Procedure: Physical therapy exercises.

INTERVENTIONS:
Procedure: Physical therapy exercises. — Exercises to treat hemiparetic cerebral palsy

SUMMARY:
This study is to investigate the effect of whole body vibration in children with hemiparetic cerebral palsy on range of motion of shoulder, elbow and wrist and muscle strength of shoulder abductors and flexors, elbow flexors and extensors, wrist extensors and flexors.

DETAILED DESCRIPTION:
Studies show efficacy of whole body vibration in reducing spasticity, improving strength, balance, ankle dorsiflexion angle and gait parameters in post stroke and spinal cord injury patients improving posture and balance in patients with Parkinson's disease and multiple sclerosis. Although research suggests a positive influence of vibration on motor performance in individuals with neurological disorders, there are very limited numbers of studies in children with cerebral palsy.

Few Studies Have Shown improvement in children with cerebral palsy: spasticity decrease as measured by isokinetic dynamometer. Strength of muscles increase as measured by hand held dynamometer. Motor function increase as measured by Gross Motor Function Measure and Gross Motor Function Classification Scale. Increase of the activation and the co- activation of biceps and triceps. Vibrations increase bone mass and muscle strength in upper limbs.

Vibration therapy decreases spasticity and improve motor performance in children with cerebral palsy. Reduce flexors spasticity and improve functions in the rehabilitation of upper limb spasticity. Focal muscle vibration on triceps brachii muscle can reduce the spasticity for both elbow and wrist joint muscles.

So in this study, the investigators are trying to implement an additional rehabilitation method for upper limbs in hemiparetic children to improve their upper limb range of motion and strength which will reflect an improvement in their upper limb functions and activities of daily living.

ELIGIBILITY:
Inclusion criteria:

Children will be included if they have the following:

1. Children diagnosed as hemiparetic cerebral palsy.
2. Children of both sexes in the age group ranging from 3 to 6 years.
3. Spasticity will be grade 1 and 1+ according to modified Ashworth scale.
4. They will be selected with Level I and II according to Gross Motor Function Classification (GMFCS).
5. Children could understand and follow commands given by the therapist.

Exclusion criteria:

Children will be excluded if they have any of the following:

1. History of convulsions and epilepsy.
2. Children with impaired cognitive function.
3. Any surgical procedure for correction of deformity or soft tissue release in the past one year.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in shoulder joint abduction range of motion. | Change from Baseline shoulder joint abduction range of motion at one month.
  Measurement of range of motion of shoulder joint abduction using the digital Goniometer.
Change in shoulder joint flexion range of motion. | Change from Baseline shoulder joint flexion range of motion at one month.
  Measurement of range of motion of shoulder joint flexion using the digital Goniometer.
Change in elbow joint flexion range of motion. | Change from Baseline elbow joint flexion range of motion at one month.
  Measurement of range of motion of elbow joint flexion using the digital Goniometer.
Change in elbow joint extension range of motion. | Change from Baseline elbow joint extension range of motion at one month.
  Measurement of range of motion of elbow joint extension using the digital Goniometer.
Change in wrist joint extension range of motion. | Change from Baseline wrist joint extension range of motion at one month.
  Measurement of range of motion of wrist joint extension using the digital Goniometer.
Change in wrist joint flexion range of motion. | Change from Baseline wrist joint flexion range of motion at one month.
  Measurement of range of motion of wrist joint flexion using the digital Goniometer.
Change in strength of shoulder abductors muscles. | Change from Baseline strength of shoulder abductors muscles at one month.
  Measurement of strength of shoulder abductors muscles using the Lafayette handheld dynamometer
Change in strength of shoulder flexors muscles. | Change from Baseline strength of shoulder flexors muscles at one month.
  Measurement of strength of shoulder flexors muscles using the Lafayette handheld dynamometer
Change in strength of elbow flexors muscles. | Change from Baseline strength of elbow flexors muscles at one month.
  Measurement of strength of elbow flexors muscles using the Lafayette handheld dynamometer
Change in strength of elbow extensors muscles. | Change from Baseline strength of elbow extensors muscles at one month.
  Measurement of strength of elbow extensors muscles using the Lafayette handheld dynamometer
Change in strength of wrist extensors muscles. | Change from Baseline strength of wrist extensors muscles at one month.
  Measurement of strength of wrist extensors muscles using the Lafayette handheld dynamometer
Change in strength of wrist flexors muscles. | Change from Baseline strength of wrist flexors muscles at one month.
  Measurement of strength of wrist flexors muscles using the Lafayette handheld dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Haytham Morsi, M.Sc., Study Director — Cairo University
Locations (1):
- Ministry of Health, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No